CLINICAL TRIAL: NCT04654312
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Influence of Hydrochlorothiazide on Dermal Photosensitivity and DNA Stability - a Pilot Study (HCTox Study)
Brief Title: Study to Evaluate the Influence of Hydrochlorothiazide on Dermal Photosensitivity and DNA Stability - a Pilot Study (HCTox Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HCTox
Record Dates: First submitted 2020-11-24; First posted 2020-12-04 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2021-07

CONDITIONS: Photosensitivity
MeSH Terms: conditions — Photosensitivity Disorders | interventions — Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: National, prospective, single-center, double-blind, parallel group, randomized, controlled, interventional Trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intake of HCT 25 mg, 1 tablet/d for 15 days
  Interventions: Drug: Hydrochlorothiazide
- Placebo (Placebo Comparator): Intake of Placebo, 1 tablet/d for 15 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrochlorothiazide — Please see arm descriptions
  Other Names: HCT
  Arms: Intervention
Drug: Placebo — Please see arm descriptions
  Arms: Placebo

SUMMARY:
The clinical trial is designed as a national, prospective, single-center, double-blind, parallel group, randomized, controlled, interventional trial to investigate whether a therapy with HCT compared with placebo can affect dermal photosensitivity and DNA stability.

DETAILED DESCRIPTION:
Previously published retrospective analyses leading to the official warning about the use of hydrochlorothiazide (HCT).

The underlying pilot study examins, if the intake of HCT leads to increased dermal photosensitivity and in combination with UV-exposition to a DNA-damage of the skin.

Up until today, there is no prospective, randomized, placebo-controlled trial investigating the impact of HCT on dermal photosensitivity in greater detail. The pilot trial is designed as feasibility study to clarify the impact of HCT on dermal photosensitivity. This may facilitate evidence-based recommendations as to whether or not HCT increases the risk for skin cancer. Of note, HCT is one of most frequently prescribed drugs in Germany.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is willing and able to participate and provides written informed consent;
2. Healthy subjects with no concomitant medical conditions;
3. Age ≥ 18 years;
4. The subject is willing to take HCT 25 mg a day although not clinically indicated;
5. The subject is willing to undergo controlled UV-exposition although not clinically indicated;
6. Skin type I - IV.

Exclusion Criteria:

1. History of any cardiac disease;
2. History of any dermatologic disease;
3. Renal insufficiency (eGFR <60 ml/min/1.73m²);
4. Intake of photosensitive substances, especially intake of HCT;
5. Frequent, above-average, UV exposition (naturally or artificially);
6. Known hypertension;
7. Known electrolyte disbalance;
8. Systolic blood pressure at baseline <100 mmHg;
9. Skin type V and VI;
10. History of severe diseases, which could endanger the safety of study participant;
11. Known unresolved history of alcohol dependency or drug abuse or any other kind of dependencies
12. Intake of any of the following medications or substances: Betablockers; nitrates; barbiturates; phenothiazines; tricyclic antidepressants; vasodilatory drugs; ACE-inhibitors; NSAIDs; salicylates; phenytoin; Insulin; oral antidiabetic drugs; vasoconstrictors; glycosides; substances lowering blood-urea levels; substances causing a Long-QT-Syndrome; chinidine; carbamazepine; cyclosporine; cholecalciferol; potassium salts; amantadine; allopurinol; methyldopa; cholestyramine; colestipol; other diuretics; lithium; cytostatic drugs;
13. Women in childbearing age and not using medically acceptable effective contraception refer to CTFG: The study population includes female of childbearing potential. Female of childbearing potential have to agree to comply with the applicable contraceptive requirements of the protocol for the duration of the study or having post-menopausal status or be permanently sterilized (at least 6 weeks post-sterilization). Highly effective contraception is defined as a contraceptive method with failure rate of less than 1 % per year when used consistently and correctly and when applicable, in accordance with the product label;
14. Subject is pregnant (e.g., positive ß-hCG test) or is breast feeding;
15. Hypersensitivity to the active substance, to HCT or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Changes in subjects´ minimal-erythema-dose (MED). | 2 weeks
  The MED is the minimal erythema dose, meaning the minimal dose of energy (in this case provided by UV-exposition) per area that leads to a clinically visible skin reaction, mainly a slight reddening.
  The MED is assessed by a clinical tool called the light-stair.
Amount of excretion of pyrimidine-dimers (PD) in urine. | 26 days
  Changes from Baseline Visit to Day 26

SECONDARY OUTCOMES:
Changes in blood-serum vitamin-D levels. | 26 days
  Changes from Baseline Visit to Day 24
Changes in blood pressure. | 26 days
  Changes from Baseline Visit to Day 24

OTHER OUTCOMES:
Changes in electrolytes (Na+, K+) | 26 days
  Changes from Baseline Visit to Day 24
Changes in kidney function (eGFR) | 26 days
  Changes from Baseline Visit to Day 24
Changes in blood count | 26 days
  Changes from Baseline Visit to Day 24

CONTACTS AND LOCATIONS:
Overall Officials: Felix Mahfoud, MD, Principal Investigator — Saarland University Hospital
Locations (1):
- Saarland University Hospital, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gotzinger F, Hohl M, Lauder L, Millenaar D, Kunz M, Meyer MR, Ukena C, Lerche CM, Philipsen PA, Reichrath J, Bohm M, Mahfoud F. A randomized, placebo-controlled, trial to assess the photosensitizing, phototoxic and carcinogenic potential of hydrochlorothiazide in healthy volunteers. J Hypertens. 2023 Nov 1;41(11):1853-1862. doi: 10.1097/HJH.0000000000003558. Epub 2023 Sep 13. PMID 37702559
- See also: Hydrochlorothiazid - Risiko von nichtmelanozytärem Hautkrebs [Basalzellkarzinom (Basaliom); Plattenepithelkarzinom der Haut (Spinaliom): Rote-Hand-Brief vom 17. Oktober 2018. — https://www.bfarm.de/SharedDocs/Risikoinformationen/Pharmakovigilanz/DE/RHB/2018/rhb-hydrochlorothiazid.html